CLINICAL TRIAL: NCT07264907
Title: Tai Chi Improves Sleep Quality in Patients With Mild to Moderate Chronic Insomnia
Brief Title: Tai Chi Improves Sleep Quality in Mild to Moderate Chronic Insomnia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025350H; 2025350H (Other: BeijingSU)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Tai Ji; Walking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention Group: If subjects are eligible to participate in this study, they will be randomly assigned by the doctor to undergo the following two phases, including a screening and baseline assessment period, an intervention period, and a follow-up period. The specific assessments conducted in each phase are as follows: The entire trial consists of 3 stages, with each stage comprising 2 periods (a test period or a control period, each lasting 1 week/2 weeks). After enrollment, patients will be randomly allocated to either the test period (Tai Chi) or the control period (walking). During the study, subjects will be required to cooperate with doctors to complete relevant questionnaires and follow-up assessments.
  Interventions: Other: Tai Chi and Walking

INTERVENTIONS:
Other: Tai Chi and Walking — 1. Frequency: Train three times a week on a fixed day (e.g., Monday, Wednesday, Friday) to avoid two consecutive days of no training and ensure continuity;
  2. Duration: 40 minutes for the basic preparation phase, and 60 minutes for the advanced learning and integration phase (including warm-up, core training, and relaxation).
  3. Attendance requirement: Participants must complete at least 19 training sessions (24 sessions over 8 weeks with an attendance rate of ≥80%). In case of absence due to special circumstances, they must complete supplementary training via online video (instructor-recorded action breakdowns) within one week, with the same duration as regular sessions.

SUMMARY:
What are the requirements for participating in this study?

1. Age 40 to 69, gender unlimited;
2. Insomnia symptoms (difficulty falling asleep, frequent awakenings during sleep, early morning awakening, etc.) occurring three or more times per week for three months or longer (meeting DSM-5 diagnostic criteria for chronic insomnia and International Classification of Sleep Disorders standards); 3.7 points <ISI baseline score ≤ 21 points (mild to moderate insomnia);

4. The patient is dissatisfied (option 3) or very dissatisfied (option 4) with their current sleep 5. The incubation period or wake time after falling asleep is more than 30 minutes, and the total sleep time is less than 6.5 hours per day; 6. Willing to follow the exercise prescription and coach's guidance, and cooperate with the exercise intervention for 6 weeks; 7. Being able to maintain consistent lifestyle and sleep patterns throughout the study; 8. Fixed residence and no expectation of moving or traveling within 6 weeks; 9. Sign the informed consent form.

You are not eligible to participate in this study if you meet any of the following criteria:

1. Exclude diseases that affect sleep (such as tumors, dementia, obstructive sleep apnea, etc.);
2. Taking medications that may affect sleep (such as steroid hormones, sleeping pills, psychotropic drugs);
3. Abuse of alcohol or drugs in the last 3 months;
4. Liver or kidney dysfunction;
5. History of severe cardiovascular and cerebrovascular diseases;
6. History of mental illness;
7. Expect to work night shifts or travel across time zones or sleep irregularly during the study period;
8. Participated in other intervention clinical trials, including drugs, nutritional preparations and medical devices, within 3 months before the study.

What will I experience if I participate in this study? If eligible, participants will be randomly assigned by physicians to one of two study phases: the screening and baseline assessment phase, or the intervention and follow-up phase. The trial consists of three phases, each containing two phases (experimental or control, lasting 1-2 weeks). After enrollment, participants will be randomly assigned to either the Tai Chi intervention group or the walking control group. Throughout the study, participants must cooperate with physicians to complete relevant questionnaires and attend scheduled follow-up visits.

What might be the benefits of participating in this study? The research team will cover all expenses for the exercise program. Participants will receive free exercise training, physiological counseling, and standardized assessments throughout the study, including follow-up sessions. Our previous sports medicine research shows that 12 weeks of Tai Chi therapy can significantly improve insomnia symptoms.

What are the risks of participating in this study? Participants who have not exercised for a long time may have adverse reactions such as muscle pain and joint pain caused by exercise in the early stage of the experiment or during the study, or even lead to the termination of the experiment.

Is participation in this study mandatory? No, participation in this study is entirely voluntary.

Can I quit the study midway? Yes, you can opt out at any time, and this will not affect your legal right to continue regular checkups or treatments.

Are my personal information confidential? Your personal privacy will be strictly protected within the bounds of applicable laws. Monitoring officers, auditors, ethics committees, and management authorities shall be permitted to directly access participants 'original medical records to verify clinical trial procedures and data, provided such access does not violate applicable laws and regulations or infringe upon participants' privacy. Throughout the study, participants have the right to withdraw from the research at any time without facing discrimination, retaliation, or disruption of medical services. All personal information collected during the study remains confidential. Participants are entitled to consult our physicians with any questions at any time.

Patient Statement (Please tick in parentheses):

1. I have reviewed the relevant research materials for this study (version v1.0)···········□
2. I have carefully considered the matter, consulted a doctor about the relevant issues, and received satisfactory answers······□
3. I understand that participation in this study is voluntary and that I have the right to withdraw from this study at any time without any reason without affecting my medical treatment and rights·····□
4. I understand that my relevant materials will be reviewed by the research unit or members of the strict management agency in this study. I agree to the above personnel reviewing and using my relevant materials. ·······················□
5. I agree to participate in this study·····························□

DETAILED DESCRIPTION:
informed consent

Please read the following carefully before you decide to participate in this study. If you are willing to participate, please fill out the informed consent form.

Insomnia, a condition marked by difficulty falling asleep or maintaining deep sleep, is characterized by persistent sleep disturbances. It often manifests alongside daytime fatigue, drowsiness, irritability, and in severe cases, depressive or anxious symptoms. Epidemiological studies indicate that 6% to 10% of adults experience insomnia, with nearly half of the population suffering from it annually. Women and older adults are particularly vulnerable. The primary treatment goals are to improve sleep quality and alleviate functional impairments caused by sleep disorders. Current approaches include psychotherapy (such as cognitive behavioral therapy, group behavioral therapy, or brief cognitive behavioral therapy) and medication (sleep aids, antidepressants, antipsychotics, and melatonin). Alternative therapies like acupuncture and herbal medicine are also used, though their clinical effectiveness remains unproven. The American Medical Association's Evidence-Based Clinical Practice Guidelines recommend cognitive behavioral therapy for chronic insomnia (strongly recommended, moderate evidence), while medication use requires careful evaluation of efficacy, side effects, and cost-effectiveness (low-quality evidence). Long-term use of sleep or psychiatric medications should only be considered for strictly defined conditions, as potential risks of dependency and adverse reactions remain a concern for both patients and clinicians.

Although traditional drug therapy can improve sleep in the short term, long-term use poses issues such as dependence and side effects, making it difficult to serve as an ideal long-term intervention. Therefore, exploring a safe, effective, and non-pharmacological intervention method has become an important direction in current insomnia treatment research. Tai Chi, as a traditional Chinese health-preserving method, integrates breathing regulation, mental guidance, and slow limb movements, emphasizing the unity of body and mind and the balance of yin and yang. Numerous studies have confirmed its positive effects in regulating the nervous system, alleviating anxiety, and improving sleep quality. Recent empirical studies both domestically and internationally have also found that regular practice of Tai Chi can effectively improve sleep quality, shorten the time to fall asleep, and prolong the deep sleep stage, particularly showing significant efficacy for middle-aged and elderly insomnia patients.

What are the requirements for participating in this study?

1. Age 40 to 69, gender unlimited;
2. Insomnia symptoms (difficulty falling asleep, frequent awakenings during sleep, early morning awakening, etc.) occurring three or more times per week for three months or longer (meeting DSM-5 diagnostic criteria for chronic insomnia and International Classification of Sleep Disorders standards); 3.7 points <ISI baseline score ≤ 21 points (mild to moderate insomnia);

4. The patient is dissatisfied (option 3) or very dissatisfied (option 4) with their current sleep 5. The incubation period or wake time after falling asleep is more than 30 minutes, and the total sleep time is less than 6.5 hours per day; 6. Willing to follow the exercise prescription and coach's guidance, and cooperate with the exercise intervention for 6 weeks; 7. Being able to maintain consistent lifestyle and sleep patterns throughout the study; 8. Fixed residence and no expectation of moving or traveling within 6 weeks; 9. Sign the informed consent form.

You are not eligible to participate in this study if you meet any of the following criteria:

1. Exclude diseases that affect sleep (such as tumors, dementia, obstructive sleep apnea, etc.);
2. Taking medications that may affect sleep (such as steroid hormones, sleeping pills, psychotropic drugs);
3. Abuse of alcohol or drugs in the last 3 months;
4. Liver or kidney dysfunction;
5. History of severe cardiovascular and cerebrovascular diseases;
6. History of mental illness;
7. Expect to work night shifts or travel across time zones or sleep irregularly during the study period;
8. Participated in other intervention clinical trials, including drugs, nutritional preparations and medical devices, within 3 months before the study.

What will I experience if I participate in this study? If eligible, participants will be randomly assigned by physicians to one of two study phases: the screening and baseline assessment phase, or the intervention and follow-up phase. The trial consists of three phases, each containing two phases (experimental or control, lasting 1-2 weeks). After enrollment, participants will be randomly assigned to either the Tai Chi intervention group or the walking control group. Throughout the study, participants must cooperate with physicians to complete relevant questionnaires and attend scheduled follow-up visits.

What might be the benefits of participating in this study? The research team will cover all expenses for the exercise program. Participants will receive free exercise training, physiological counseling, and standardized assessments throughout the study, including follow-up sessions. Our previous sports medicine research shows that 12 weeks of Tai Chi therapy can significantly improve insomnia symptoms.

What are the risks of participating in this study? Participants who have not exercised for a long time may have adverse reactions such as muscle pain and joint pain caused by exercise in the early stage of the experiment or during the study, or even lead to the termination of the experiment.

Is participation in this study mandatory? No, participation in this study is entirely voluntary.

Can I quit the study midway? Yes, you can opt out at any time, and this will not affect your legal right to continue regular checkups or treatments.

Are my personal information confidential? Your personal privacy will be strictly protected within the bounds of applicable laws. Monitoring officers, auditors, ethics committees, and management authorities shall be permitted to directly access participants 'original medical records to verify clinical trial procedures and data, provided such access does not violate applicable laws and regulations or infringe upon participants' privacy. Throughout the study, participants have the right to withdraw from the research at any time without facing discrimination, retaliation, or disruption of medical services. All personal information collected during the study remains confidential. Participants are entitled to consult our physicians with any questions at any time.

Patient Statement (Please tick in parentheses):

1. I have reviewed the relevant research materials for this study (version v1.0)···········□
2. I have carefully considered the matter, consulted a doctor about the relevant issues, and received satisfactory answers······□
3. I understand that participation in this study is voluntary and that I have the right to withdraw from this study at any time without any reason without affecting my medical treatment and rights·····□
4. I understand that my relevant materials will be reviewed by the research unit or members of the strict management agency in this study. I agree to the above personnel reviewing and using my relevant materials. ·······················□
5. I agree to participate in this study·····························□

Subject signature:

Signature of authorized agent: Relationship with subject: Signature of authorized agent: Relationship with subject:

Contact: Date: Contact: Date:

The researchers stated:

I have carefully explained to the subject the nature of the study and the benefits and risks of participating in it. His signature is valid. Medical problems, language or educational level do not prevent him from understanding the above.

Researcher signature:

Contact: Date: Contact: Date:

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 69, gender unlimited;
2. Insomnia symptoms (difficulty falling asleep, frequent awakenings during sleep, early morning awakening, etc.) occurring three or more times per week for three months or longer (meeting DSM-5 diagnostic criteria for chronic insomnia and International Classification of Sleep Disorders standards); 3.7 points <ISI baseline score ≤ 21 points (mild to moderate insomnia);

4. The patient is dissatisfied (option 3) or very dissatisfied (option 4) with their current sleep 5. The incubation period or wake time after falling asleep is more than 30 minutes, and the total sleep time is less than 6.5 hours per day; 6. Willing to follow the exercise prescription and coach's guidance, and cooperate with the exercise intervention for 6 weeks; 7. Being able to maintain consistent lifestyle and sleep patterns throughout the study; 8. Fixed residence and no expectation of moving or traveling within 6 weeks; 9. Sign the informed consent form.

Exclusion Criteria:

1. Exclude diseases that affect sleep (such as tumors, dementia, obstructive sleep apnea, etc.);
2. Taking medications that may affect sleep (such as steroid hormones, sleeping pills, psychotropic drugs);
3. Abuse of alcohol or drugs in the last 3 months;
4. Liver or kidney dysfunction;
5. History of severe cardiovascular and cerebrovascular diseases;
6. History of mental illness;
7. Expect to work night shifts or travel across time zones or sleep irregularly during the study period;
8. Participated in other intervention clinical trials, including drugs, nutritional preparations and medical devices, within 3 months before the study.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he study population consists of individuals aged 40 to 69 years diagnosed with insomnia, defined according to the diagnostic criteria of the International Classification of Sleep Disorders (ICSD-3) or the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Eligible participants typically report persistent sleep disturbances (e.g., difficulty falling asleep, frequent nighttime awakenings, early-morning awakening, or non-restorative sleep) lasting at least 3 months, occurring at least 3 nights per week, and causing significant daytime impairment (such as fatigue, mood disturbances, cognitive dysfunction, or reduced work/activity capacity).
  This age group (40-69 years) is characterized by a high prevalence of insomnia, often associated with physiological changes (e.g., declining sleep efficiency, altered circadian rhythms), chronic comorbidities (e.g., hypertension, diabetes, musculoskeletal disorders), psychological stress, or lifestyle factors (e.g., sedentary behavior, irreg
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire designed to assess subjective sleep quality over a 1-month period. Developed by Buysse et al. in 1989, it consists of 19 individual items categorized into 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored on a 0-3 scale, with total scores ranging from 0 to 21. A total score ≥ 7 indicates poor sleep quality, while a score < 7 reflects good sleep quality.
  The PSQI is recognized for its simplicity, reliability, and validity across diverse populations, including healthy individuals, patients with chronic diseases, and those with sleep disorders. It is extensively employed in clinical research, epidemiological studies, and clinical practice to evaluate sleep outcomes, particularly in fields such as medicine, psychology, public health, and complementary and altern